CLINICAL TRIAL: NCT05472857
Title: Clinical Study of CLDN18.2-targeting Chimeric Antigen Receptor-modified Autologous T Cells in Advanced Solid Tumors With Positive CLDN18.2 Expression
Brief Title: Clinical Study of CLDN18.2-targeting CAR T Cells in Advanced Solid Tumors With Positive CLDN18.2 Expression
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Immunofoco Biotechnology Co., Ltd (Industry)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMC002-CT01
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Advanced Ovarian Carcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Claudin 18.2 CAR-T
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Accelerated titration and Bayesian optimal interval design (BION) dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-claudin18.2 chimeric antigen receptor T-cell therapy (Experimental): anti-claudin18.2 chimeric antigen receptor T-cell therapy，infusion
  Interventions: Biological: Claudin 18.2 CAR-T

INTERVENTIONS:
Biological: Claudin 18.2 CAR-T — treatment with anti-claudin18.2 chimeric antigen receptor T-cell infusion
  Other Names: IMC002

SUMMARY:
This is an open label, multi-center, Phase 1 clinical trial to evaluate the safety and efficacy of autologous claudin18.2 chimeric antigen receptor T-cell therapy in advanced solid tumors with positive CLDN18.2 expression

DETAILED DESCRIPTION:
Following consent, patients must have tumor tissue evaluated by CLDN18.2 IHC assay. Patients meeting all eligibility criteria will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (IMC002). Following manufacture of the drug product, subjects will receive preconditioning prior to IMC002 infusion. All subjects will be asked to continue to undergo long-term gene safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for screening for potential inclusion in the study:

  1. The age is between 18 and 70 years old (including the boundary value), both male and female.
  2. Subjects with advanced CLDN 18.2 positive malignant solid tumors confirmed by histology or cytology in the past (including advanced gastric cancer or esophagogastric junction adenocarcinoma, advanced pancreatic cancer, and metastatic ovarian cancer without standard treatment).
  3. All subjects are required to provide tumor tissue specimens that can be used for CLDN 18.2 analysis, which must be tumor histopathological specimens within 24 months before signing the informed consent, or fresh biopsy specimens collected within 6 months before cell reinfusion ; CLDN 18.2 histological staining of biopsy tumor tissue specimens is positive (defined as staining intensity ≥ 1+, positive rate ≥ 10%), the recommended antibody for detection is: Anti-Claudin18.2 antibody.
  4. Estimated life expectancy≥12 weeks.
  5. At least 1 measurable lesion per RECIST version1.1;
  6. ECOG performance status score of 0-1.
  7. The subject has adequate organ and bone marrow function.
  8. All toxic reactions caused by previous anti-tumor therapy were relieved to grade 0-1 (according to NCI CTCAE version 5.0) or to an acceptable level for inclusion/exclusion criteria.
  9. Fertility status: Female patients of childbearing age or male patients whose sexual partners are females of childbearing age are willing to take medically approved high-efficiency contraceptive measures such as intrauterine devices from the time of signing the informed consent to 6 months after the last cell infusion or condoms (women of childbearing age include premenopausal women and women within 24 months of postmenopause).
  10. Subjects must sign and date written informed consent.
  11. Subjects must be voluntary and able to comply with predetermined treatment regimens, laboratory tests, follow-up and other research requirements.

Exclusion Criteria:

* Subjects who meet any of the following conditions are not eligible for this study;

  1. Pregnant and lactating women.
  2. Known history of human immunodeficiency virus (HIV) infection; acute or chronic active hepatitis B (HBsAg positive or HBsAb positive, and HBV-DNA positive); acute or chronic active hepatitis C (HCV antibody positive) , and HCV-RNA was positive). Syphilis antibody positive; EB virus DNA quantification >500 copies (or according to the positive standard detected by each research center); cytomegalovirus (CMV) infection (IgM positive).
  3. Serious infection in active stage or poorly controlled clinically.
  4. There is currently a heart disease requiring treatment or hypertension that is poorly controlled by the investigator (defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure > 90 mmHg after standardized antihypertensive drug treatment).
  5. Within 6 months before cell reinfusion, any of the following cardiac clinical symptoms or diseases: left ventricular ejection fraction (LVEF) < 50%; previous history of coronary heart disease, myocardial infarction, severe heart failure and severe arrhythmia.
  6. Evidence of major coagulation disorder or other significant bleeding risk: including but not limited to receiving conventional anticoagulation therapy (such as warfarin or heparin). Patients require long-term antiplatelet therapy (aspirin, dose >300mg/day; clopidogrel, dose >75mg/day); dipyridamole, ticlopidine or cilostazol, etc.
  7. Subjects requiring systemic therapy with corticosteroids or other immunosuppressive drugs during the treatment period.
  8. Blood oxygen saturation ≤95% before treatment (refers to pulse oxygen detection).
  9. Diffuse lung metastases.
  10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis, and symptomatic interstitial lung disease or active pneumonia found on chest CT scan within 4 weeks before the first study drug treatment.
  11. Uncontrollable pleural effusion, pericardial effusion and ascites effusion existed before enrollment.
  12. Poorly controlled diabetes (glycated hemoglobin HbA1c ≥ 8%).
  13. Received systemic steroids equivalent to >15mg/day prednisone within 2 weeks before apheresis, except inhaled steroids.
  14. The subject has developed new arrhythmias, including but not limited to uncontrolled arrhythmias, hypotension requiring vasopressors, bacterial, fungal or viral infections requiring intravenous antibiotics prior to preconditioning . Subjects using the trial antibiotic to prevent infection were at the discretion of the investigator to continue participating in the trial.
  15. Known past or current hepatic encephalopathy requiring treatment; patients with current or history of central nervous system disease; central nervous system metastases or meningeal metastases with clinical symptoms, or other evidence of central nervous system metastases or Meningeal metastases have not yet been controlled, and were judged by the investigator to be unsuitable for enrollment.
  16. Patients with previous or concomitant malignancies, with the following exceptions: Adequately treated basal cell or squamous cell carcinoma, cured cervical or breast carcinoma in situ, primary malignancy that has been completely resected and complete remission for ≥5 years.
  17. Received other CAR-T therapy and TCR-T therapy in the past.
  18. Received the following treatments or drugs before cell reinfusion: within 28 days before cell reinfusion, received chemotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments (treatments that met the requirements of the plan before reinfusion, such as bridging therapy) Except for), or any unmarketed experimental drug treatment; received traditional Chinese medicine treatment with anti-tumor indications within 2 weeks before cell reinfusion.
  19. Subjects who have received other gene therapy in the past.
  20. Subjects with severe mental disorders.
  21. Participated in other clinical studies within the past 1 month.
  22. The investigator assesses that the subject is unable or unwilling to comply with the requirements of the research protocol.
  23. Subjects withdrew from the study for various reasons and could not participate in the study again.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | day1 - month12
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs)
Identification of Maximum Tolerated Dose (MTD) | day1 - day28
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Objective Response Rate (ORR)，as assessed by Investigators | day1 - month12
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Duration of response (DOR)，as assessed by Investigators | day1 - month12
  Duration of response (DOR) is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Disease control rate (DCR), as assessed by Investigators | day1 - month12
  Disease control rate (DCR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.
Progression-free survival (PFS), as assessed by Investigators | day1 - month12
  Progression-free survival (PFS) was defined as the time from the date of first infusion of CT041 to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Tianhang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No